CLINICAL TRIAL: NCT02146729
Title: Treatment of Thoracolumbar Spine Fractures: Percutaneously Placed Pedicle Screws Versus Open Treatment
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Research personnel changes prevented study initiation and enrollment
Sponsor: Daniel Altman (Other)
Responsible Party: Sponsor-Investigator, Daniel Altman, Orthopaedic Surgeon, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Organization: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC 5903
Record Dates: First submitted 2014-05-15; First posted 2014-05-26 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Thoracolumbar Spine Trauma
Keywords: Randomized; Thoracolumbar fractures; Spine Trauma; Percutaneous Pedicle Screw Fixation; Functional Outcome
MeSH Terms: interventions — Open Abdomen Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Percutaneous Pedicle Screw Fixation (Experimental): Percutaneous Pedicle Screw Fixation
  Interventions: Procedure: Percutaneous Pedicle Screw Fixation
- Open Treatment (Active Comparator): Midline posterior incision with instrumentation.
  Interventions: Procedure: Open Treatment

INTERVENTIONS:
Procedure: Percutaneous Pedicle Screw Fixation — Percutaneous Pedicle Screw Fixation
  Arms: Percutaneous Pedicle Screw Fixation
Procedure: Open Treatment — Midline posterior incision with instrumentation.
  Arms: Open Treatment

SUMMARY:
In patients presenting with Type A and Type B1, B2 thoracolumbar fractures, there is a lack of evidence demonstrating similar outcomes between patients treated with percutaneous pedicle screws and those treated openly. It has been demonstrated that percutaneous pedicle screw fixation has fared well for patients in the short term; however, it is unclear whether the outcomes are equivalent or inferior/superior compared to open treatment.

The authors seek to establish a high-level evidence base to determine clinical patient outcomes, radiographic outcomes, as well as cost-effectiveness data in comparing thoracolumbar burst fracture patients treated with percutaneous pedicle screws, open treatment, and brace treatment. Additionally, the authors seek to establish data relating to patient occupational data, complications, and need for further surgery (revision/removal of hardware), as well as short-term variables relating to hospital visit (length of stay, estimated blood loss, time under fluoroscopy).

ELIGIBILITY:
Inclusion Criteria:

* All patients from ages 18 and older who present to Allegheny General Hospital with an acute thoracolumbar fracture will be considered eligible for the study (i.e. <3 weeks from trauma date).
* Minor fractures around the fracture site or compression fractures will be permitted if they do not require treatment
* For the purposes of the study, patients must be English-speaking and live within the 100 mile radius from the greater Pittsburgh area for consent and follow-up purposes
* Patients who cannot safely undergo brace treatment due to comorbidities such as obesity, pulmonary injury, elderly status, reliability, and multitrauma
* Patients must have Type A or Type B1,B2 thoracolumbar fracture (must be able to correct deformity through percutaneous instrumentation)

Exclusion Criteria:

* Patients presenting with a neurologic deficit
* Patients who receive a laminectomy for decompression of the neural elements
* Patients who have a significant head injury
* Oncologic patients
* Women who were found to be pregnant or breast feeding at any point during their admission, hospital stay, treatment, or clinical follow-up.
* Individuals who are currently incarcerated.
* Adolescents under 18 years of age.
* Patients who have a relative contraindication to operative treatment will be excluded - infection, skin disease, bleeding disorder, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Health Related Quality of Life Measure Scores | 24 months
  Oswestry Disability Index, Roland Morris Disability Score, Visual Analog Spine Score, Euroqol 5D-5L

SECONDARY OUTCOMES:
Radiographic Evaluations | 24 months
  Kyphosis
Cost Effectiveness | Duration of Hospital Stay (expected duration average 1 week)
Complication rate/Adverse event | 24 months
Additional medical procedures | 24 months
  Any additional medical procedures outside of the index surgery.
Length of Hospital Stay | Duration of hospital stay (expected duration average 1 week)
Estimated Blood Loss | Duration of hospital visit (expected duration- average 1 week)
  Estimated blood loss, operating time, fluoroscopy time
Return to work | 24 months
Radiographic Evaluation | 24 months
  Loss of height
Operating Time | Duration of hospital visit (expected duration 1 week)
  The time it takes to complete the index surgery from start to finish.
Fluoroscopy time | Duration of hospital stay (expected duration average 1 week)
  Duration of time the fluoroscopy was in use during the index surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Allegheny General Hospital, Department or Orthopaedic Surgery, Pittsburgh, Pennsylvania, United States